CLINICAL TRIAL: NCT01441206
Title: Safety and Pharmacokinetics of Single and Multiple Dose Rifampin in Infants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study to be redesigned.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-2314; 1K23HD068497-01 (NIH)
Record Dates: First submitted 2011-09-19; First posted 2011-09-27 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Infection
Keywords: rifampin; infants
MeSH Terms: conditions — Infections | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rifampin (Other): Cohort 1 will include infants who will be receiving up to 4 doses rifampin per study protocol.
  Interventions: Drug: rifampin
- rifampin per standard of care (No Intervention): Cohort 2: Receiving rifampin per standard of care

INTERVENTIONS:
Drug: rifampin — Infants who will be receiving up to 4 doses of rifampin per protocol(Cohort 1)
  Cohort 1:
  Dosing will be as follows:
  GA at birth < 32 weeks - PNA < 14 days: 10 mg/kg QD GA at birth < 32 weeks - PNA ≥ 14 days: 15 mg/kg QD GA at birth ≥ 32 weeks - PNA < 14 days: 15 mg/kg QD GA at birth ≥ 32 weeks - PNA ≥ 14 days: 20 mg/kg QD
  Arms: rifampin

SUMMARY:
The purpose of this study is to learn more about the safety and dosing of rifampin in infants.

DETAILED DESCRIPTION:
Pharmacokinetics and safety of rifampin will be studied in term and preterm infants who are receiving rifampin per standard of care.

ELIGIBILITY:
Cohort 1:

* Suspected systemic infection
* Infant < 121 days of age at the time of 1st dose of rifampin administration
* Sufficient intravascular access (either peripheral or central) to receive rifampin.

Cohort 2:

* Receiving rifampin per local standard of care.
* Infant < 121 days of age at the time of 1st dose of rifampin administration

Exclusion Criteria:

Cohort 1:

* History of allergic reactions to rifampin
* Aspartate aminotransferase (AST) greater than 3 times upper limit of normal
* Alanine aminotransferase (ALT) greater than 3 times upper limit of normal
* Serum creatinine greater than 1.7 mg.dL
* Urine output < 0.5 mL/hr/kg over the prior 24 hours
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study

Cohort 2:

* None

Max Age: 121 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve 0-24 hours for rifampin | Sampling for 24 hr dosing:Dose 1:0-15min,30-60min,1-3hr,3-6hr, 6-12hr,12-18hr. Dose 2,3 or 4:<15min prior to dose, 48-72hrs. Sampling for 12 hr dosing:Dose 1: 0-15min, 0.5-1hr, 1-2hr, 2-4hr, 5-8hr, 8-10 hr. Dose 2, 3 or 4:<15min prior to dose, 24-36hr
Peak plasma concentration of rifampin | Sampling for 24 hr dosing:Dose 1:0-15min,30-60min,1-3hr,3-6hr, 6-12hr,12-18hr. Dose 2,3 or 4:<15min prior to dose, 48-72hrs. Sampling for 12 hr dosing:Dose 1: 0-15min, 0.5-1hr, 1-2hr, 2-4hr, 5-8hr, 8-10 hr. Dose 2, 3 or 4:<15min prior to dose, 24-36hr
Clearance of rifampin | Sampling for 24 hr dosing:Dose 1:0-15min,30-60min,1-3hr,3-6hr, 6-12hr,12-18hr. Dose 2,3 or 4:<15min prior to dose, 48-72hrs. Sampling for 12 hr dosing:Dose 1: 0-15min, 0.5-1hr, 1-2hr, 2-4hr, 5-8hr, 8-10 hr. Dose 2, 3 or 4:<15min prior to dose, 24-36hr
Volume of distribution at steady state | Sampling for 24 hr dosing:Dose 1:0-15min,30-60min,1-3hr,3-6hr, 6-12hr,12-18hr. Dose 2,3 or 4:<15min prior to dose, 48-72hrs. Sampling for 12 hr dosing:Dose 1: 0-15min, 0.5-1hr, 1-2hr, 2-4hr, 5-8hr, 8-10 hr. Dose 2, 3 or 4:<15min prior to dose, 24-36hr
Half life of rifampin | Sampling for 24 hr dosing:Dose 1:0-15min,30-60min,1-3hr,3-6hr, 6-12hr,12-18hr. Dose 2,3 or 4:<15min prior to dose, 48-72hrs. Sampling for 12 hr dosing:Dose 1: 0-15min, 0.5-1hr, 1-2hr, 2-4hr, 5-8hr, 8-10 hr. Dose 2, 3 or 4:<15min prior to dose, 24-36hr

SECONDARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability. | From the time of the first dose to 3 days after the last dose; serious adverse events will be collected from the first dose of rifampin to 7 days after the last dose of rifampin.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M. Laughon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States